CLINICAL TRIAL: NCT06917599
Title: Effect Of Low-Level Laser Therapy Versus Saline On Wound Healing Of Primary Molars Extraction: A Randomized Clinical Trial
Brief Title: Low-Level Laser Therapy vs. Saline for Wound Healing After Primary Molar Extraction.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Mostafa Kamel Sallem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLLT25
Record Dates: First submitted 2025-03-23; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Wound-healing
Keywords: laser; therapy; low-level; wound healing; molar; extraction; oral
MeSH Terms: interventions — Low-Level Light Therapy; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-level laser therapy (Experimental): Effect of Low-level laser therapy in wound healing after primary molar extraction
  Interventions: Device: Low-level laser
- Saline (Active Comparator): Normal saline in wound healing after primary molar extraction
  Interventions: Other: Saline Solution (NaCl 0,9%)

INTERVENTIONS:
Device: Low-level laser — Effect of Low-level laser therapy in wound healing after primary molar extraction
  Arms: Low-level laser therapy
Other: Saline Solution (NaCl 0,9%) — Following the extraction, a piece of gauze soaked in normal saline solution (NSS) will be placed over the socket. Both parents and children will be instructed to keep the gauze in place for 45 minutes
  Arms: Saline

SUMMARY:
To evaluate the effect of low level laser therapy versus the saline on wound healing after extraction of primary Molars

ELIGIBILITY:
Inclusion Criteria:

* ● Children aged from 4 to 6 years.

  * Children of both genders.
  * Medically fit ASA I.
  * Children with badly decayed primary molars beyond repair and indicated for extraction.
  * Parents acceptance to participate in the study.
  * Cooperative children.
  * Antibiotics and painkillers have been stopped at least 12 hours prior to the procedure.(Özer et al., 2024)
  * Teeth with at least two-thirds of the root.

Exclusion Criteria:

* ● Uncooperative children.

  * Lack of informed consent by the child patient's parent to be approved ethically.
  * Unable to attend follow-up visits to avoid attrition bias by decreasing the number of drop off cases.
  * Medical history includes conditions such as prolonged bleeding, platelet disorders, hypersensitivity, allergic reactions to pain relievers, contraindications to laser therapy, and acute pain.
  * Teeth with root lengths less than two-third of the normal root length or those who experienced extensive iatrogenic trauma during tooth extraction.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Presence of granulation tissue | Follow-up day of, 3 days and 7 days after extraction
  binary outcome will be recorded by clinical examination as presence or absence of granulation tissue using Landry, Turnbull, Howley Index

SECONDARY OUTCOMES:
Assessment of tissue color | Follow-up day of, 3 days, and 7 days after extraction
  Binary (>50% gingiva red, >25% but < 50%gingiva red, <25% gingiva red, All tissue pink) will be recorded by Clinical examination using Landry, Turnbull, and Howley Index
Rate of bleeding on palpation | Follow-up day of, 3 days, and 7 days after extraction
Presence of suppuration | Follow-up day of, 3 days, and 7 days after extraction
  Clinical examination using Landry, Turnbull, and Howley Index. Unit of measurement is binary (present /absent)
Assessment of gingival margin status | Follow-up day of, 3 days, and 7 days after extraction
Size of wound | Follow-up day of, 3 days, and 7 days after extraction
Rate of post operative pain | Follow-up day of, 3 days, and 7 days after extraction
  Score (0-10) will be recorded by Wong-Baker Pain Scale

IPD SHARING:
Plan to Share IPD: Undecided